CLINICAL TRIAL: NCT07294157
Title: Comparison of the Effects of Rest Splints and High-Intensity Laser Therapy on Pain, Function, Nerve Conduction Studies, and Grip Strength in Patients With Carpal Tunnel Syndrome
Brief Title: Comparison of Rest Splints vs High-Intensity Laser Therapy in Carpal Tunnel Syndrome
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Afyonkarahisar Health Sciences University (Other)
Responsible Party: Principal Investigator, Ramazan Tuncer, med.doctor, Afyonkarahisar Health Sciences University
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2024-KAEK-09
Record Dates: First submitted 2025-12-07; First posted 2025-12-19 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2026-01

CONDITIONS: Carpal Tunnel Syndrome (CTS)
Keywords: Carpal Tunnel Syndrome; Physical Therapy Modalities; Electromyography veya Nerve Conduction
MeSH Terms: conditions — Carpal Tunnel Syndrome

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Experimental: 1. Group (rest splint group) (Experimental): The physical therapy program we routinely provide to patients with carpal tunnel syndrome in our physical therapy unit (wrist ROM isometric strengthening, intrinsic muscle strengthening, wrist stretching, desensitization exercises, tendon gliding exercises, median nerve gliding exercises, wrist flexion and extension exercises, grip strengthening exercises) will be provided to patients with carpal tunnel syndrome in our physical therapy unit. Patients will be instructed to use a splint for rest as much as possible during the day and for as long as possible at night for a period of 6 weeks.
  Interventions: Device: Rest splint group
- Experimental: Group 2 (high-intensity laser therapy (HILT)) (Experimental): This group will receive high-intensity laser therapy applied over the carpal tunnel region. HILT delivers deep tissue photothermal and photomechanical effects, promoting tissue repair and reducing inflammation. The treatment is expected to decrease pain and improve nerve conduction and grip strength.
  Interventions: Device: high-intensity laser therapy (HILT)
- Sham Comparator: Group 3 (sham high-intensity laser therapy (HILT) ) (Sham Comparator): Participants in this group will undergo a placebo laser treatment using the same device without active laser emission. The procedure will mimic the real HILT application to ensure blinding. This group will help distinguish the true therapeutic effects of HILT from placebo responses.
  Interventions: Device: sham high-intensity laser therapy (HILT)

INTERVENTIONS:
Device: Rest splint group — We routinely provide the following physical therapy program to patients with carpal tunnel syndrome in our physical therapy unit: hand wrist ROM isometric strengthening, intrinsic muscle strengthening, hand wrist stretching, desensitization exercises, tendon gliding exercises, median nerve gliding exercises, wrist flexion and extension exercises, grip strengthening exercises) will be provided to patients with carpal tunnel syndrome in our physical therapy unit, and they will be instructed to use the resting splint as much as possible during the day and maximally at night for 6 weeks. Rest splint: The WingMed brand splint is specially designed to hold the wrist in a neutral position with volar support, allowing pronation and supination of the wrist but not allowing flexion, extension, radial, or ulnar deviation.
  Arms: Experimental: 1. Group (rest splint group)
Device: high-intensity laser therapy (HILT) — Group 2 (high-intensity laser therapy (HILT)) will undergo pulsed laser therapy using the HIRO 3 device (ASA Laser, Arcugnano, Italy) five times a week for 6 weeks (a total of 30 sessions, one session per day) in addition to the physical therapy program. During each session, a three-phase treatment program will be administered to patients once a day, accompanied by a physical therapist, consisting of nerve/tendon gliding exercises.
  Arms: Experimental: Group 2 (high-intensity laser therapy (HILT))
Device: sham high-intensity laser therapy (HILT) — The sham-HILT group will receive sham laser therapy using the HIRO 3 device (ASA Laser, Arcugnano, Italy) five times a week for six weeks (a total of 30 sessions, one session per day) in addition to the physical therapy program. After patients see that the device is turned on during the sham application, the same treatment will be applied to the same treatment area for the same duration without allowing laser current output from the device.
  Arms: Sham Comparator: Group 3 (sham high-intensity laser therapy (HILT) )

SUMMARY:
The aim of this study is to compare the effectiveness of rest splints and high-intensity laser therapy(HILT) added to physical therapy programs for patients with carpal tunnel syndrome in terms of pain, function, nerve conduction studies, and grip strength.

DETAILED DESCRIPTION:
Carpal tunnel syndrome (CTS) is the most common entrapment nerve compression, causing numbness and tingling in the hand, atrophy and muscle weakness in advanced stages. Any condition that increases the volume of the carpal tunnel and narrows the diameter of the tunnel can increase the compression of the median nerve under the transverse carpal ligament and cause symptoms. The use of a wrist splint or wrist brace is a common method of non-surgical treatment of carpal tunnel syndrome. The wrist splint is designed to allow rotation and supination, while eliminating the possibility of extension, flexion and radial-ulnar deviation.High-intensity laser therapy is used to provide symptomatic relief and reduce pain-related inflammation. The soothing effect of the laser is remarkable, especially in acute cases, but in the case of chronic disorders, the pain may be aggravated after the first treatments and is continued only if it decreases.

This study was designed as a prospective randomised controlled trial. Participants were randomised into 3 groups. The 1st group will receive wrist range of motion exercises, isometric strengthening, intrinsic muscle strengthening, wrist stretching, desensitization exercises, tendon sliding exercises, median nerve sliding exercises, wrist flexion and extension exercises, grip strengthening exercises and resting splint application for 6 weeks, 5 days a week, 30 sessions in total. The 2nd group (HILT group) will be given high intensity laser therapy 5 days a week for 6 weeks (30 sessions in total) in addition to the physical therapy program. The 3rd group will be the sham HILT group and physical therapy exercises will be applied like the other groups.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18-75 years who have been diagnosed with carpal tunnel syndrome based on their medical history, physical examination, clinical findings, and electromyography(EMG) results, who have applied to the outpatient clinic for physical therapy, and who have no contraindications for treatment will be included in the study after obtaining their consent.

Exclusion Criteria:

* Diabetes Mellitus
* Hypothyroidism
* Acromegaly
* Rheumatic Diseases
* Polyneuropathy
* Ipsilateral brachial plexopathy and traumatic nerve injury in the upper extremity
* Previous injection into the carpal tunnel within the last 6 months and physical therapy
* Pregnancy
* History of malignant tumors
* Patients with cochlear implants
* Acquired Immunodeficiency Syndrome
* History of neck and/or shoulder surgery
* Corticosteroid consumption, analgesic medication use
* Epilepsy
* Skin lesion

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Estimated)
Dates: Start 2025-12-15 (Actual); Primary Completion 2026-07-15 (Estimated); Study Completion 2026-09-15 (Estimated)

PRIMARY OUTCOMES:
Visual Analog Scale (VAS): | Baseline(pre-treatment,after 6 weeks(post treatment)-after 12 weeks(post treatment)
  Patients' musculoskeletal pain intensity was assessed using the visual analog scale (VAS). The meanings of the numbers placed on a 10 cm line from 0 to 10 were explained to the patients. It was explained that no pain was 0, the most severe pain ever experienced was 10, and moderate pain was 5 points. Based on these explanations, patients were asked to rate their pain levels for the past week.

SECONDARY OUTCOMES:
Boston Carpal Tunnel Questionnaire: | Baseline(pre-treatment,after 6 weeks(post treatment)-after 12 weeks(post treatment)
  This questionnaire determines the severity of CTS-specific symptoms and functional outcome using a scale for each. The symptom severity subgroup is determined using 11 questions scored from 1 to 5, with a maximum score of 55. The higher the score, the greater the symptom severity. The functional subgroup assesses the difficulty of 8 functional activities scored from 1 to 5, with a maximum score of 40. The higher the score, the poorer the functional capacity.
LANSS neuropathic pain assessment scale | Baseline(pre-treatment,after 6 weeks(post treatment)-after 12 weeks(post treatment)
  The Self-Rating of Neuropathic Symptoms and Signs (S-LANSS) scale will be administered to all patients to determine the presence of neuropathic pain. The SLANSS scale is a measure used to distinguish neuropathic pain from nociceptive pain. Unlike the LANSS scale, the physician does not examine the patient in this scale, making it easier to administer. The S-LANSS scale consists of a total of 7 questions. The patient fills out this scale themselves. The first 5 questions consist of questions that inquire about pain symptoms, while the last 2 questions include a clinical examination that the patient performs on themselves. The answers to the questions are yes/no. Each question has a different score. The total score on the scale is 24. A total score of 12 or higher suggests neuropathic pain. The Turkish version of the S-LANSS scale has been validated and is reliable.
Pittsburgh Sleep Quality Index (PSQI) | Baseline(pre-treatment,after 6 weeks(post treatment)-after 12 weeks(post treatment)
  This scale, used to assess sleep quality, consists of 24 questions that inquire about sleep quality over the past 4 weeks. The scale has 7 components, each of which is scored on a scale of 0-3. The total PUKİ score ranges from 0 to 21, with a score higher than 5 indicating poor sleep quality. Turkish validity and reliability studies have been conducted.
Quick DASH Questionnaire | Baseline(pre-treatment,after 6 weeks(post treatment)-after 12 weeks(post treatment)
  Created to assess functional status and symptoms by focusing on physical function in the upper extremities. This questionnaire contains a total of 11 items. Symptoms or difficulty are rated on a scale of 1 to 5. At least 10 questions must be answered to calculate the Quick DASH score. The calculation result is rated between 0 and 100.0. 0 indicates no difficulty or symptoms, while 100 indicates no activity or severe symptom
Median nerve distal motor latency | Baseline(pre-treatment,after 6 weeks(post treatment)-after 12 weeks(post treatment)
  The compound muscle action potential amplitude (CMAP) will be obtained via surface electrodes placed on the abductor pollicis brevis muscle. The active recording electrode will be placed on the muscle belly and the reference electrode on the tendon insertion. The median nerve will be stimulated 8 cm proximal to the active recording electrode. Distal motor latencies will be measured from the onset of the stimulus artifact to the onset of the CMAP.
Median nerve compound muscle action potential amplitude (CMAP) | Baseline(pre-treatment,after 6 weeks(post treatment)-after 12 weeks(post treatment)
  CMAPs will be obtained via surface electrodes placed on the abductor pollicis brevis muscle. The active recording electrode will be placed on the muscle belly, and the reference electrode will be placed at the tendon insertion. The median nerve will be stimulated 8 cm proximal to the active recording electrode. The amplitude of the CMAP will be measured from the baseline to the negative peak.
Motor nerve conduction velocity | Baseline(pre-treatment,after 6 weeks(post treatment)-after 12 weeks(post treatment)
  The compound muscle action potential amplitude (CMAP) will be obtained via surface electrodes placed on the abductor pollicis brevis muscle. The median nerves will be stimulated at the wrist and antecubital fossa levels. Distal motor latencies will be measured from the onset of the stimulus artifact to the onset of the CMAP. Motor nerve conduction velocity will be calculated by dividing the distance by the distal motor latency.
Second finger sensory nerve action potential amplitude | Baseline(pre-treatment,after 6 weeks(post treatment)-after 12 weeks(post treatment)
  Sensory nerve action potential amplitudes (SNAP) will be obtained using the orthodromic method and recorded with the second ring electrodes. The median nerves will be stimulated at the proximal and distal interphalangeal joints of the index finger and palm. Distal sensory latencies will be measured from the onset of the stimulus artifact to the onset of the SNAP.
Median nerve distal sensory latency | Baseline(pre-treatment,after 6 weeks(post treatment)-after 12 weeks(post treatment)
  Sensory nerve action potential amplitudes (SNAP) will be obtained using an orthodromic method and recorded using surface electrodes placed on the wrist. The median nerves will be stimulated at the proximal and distal interphalangeal joints of the index finger. Distal sensory latencies will be measured from the onset of the stimulus artifact to the onset of the SNAP. Sensory nerve conduction velocity will be calculated by dividing the distance by the distal sensory latency.
)Sensory nerve conduction velocity | Baseline(pre-treatment,after 6 weeks(post treatment)-after 12 weeks(post treatment)
  Sensory nerve action potential amplitudes (SNAP) will be obtained using an orthodromic method and recorded with ring electrodes. The median nerves will be stimulated at the proximal and distal interphalangeal joints of the index finger. Distal sensory latencies will be measured from the onset of the stimulus artifact to the onset of the SNAP. Sensory nerve conduction velocity will be calculated by dividing the distance by the distal sensory latency.
Grip strength | Baseline(pre-treatment,after 6 weeks(post treatment)-after 12 weeks(post treatment)
  A hand dynamometer (JAMAR) will be used to assess grip strength. The patient will perform three consecutive tests while sitting with shoulders abducted and neutrally rotated, elbow flexed at 90°, and forearm and wrist in a neutral position. The best of these measurements will be recorded in kilograms.
Pinchmeter | Baseline(pre-treatment,after 6 weeks(post treatment)-after 12 weeks(post treatment)
  A pinchmeter will be used to evaluate pulp-to-pulp grip strength. The patient will sit with shoulders abducted and neutrally rotated, elbow flexed at 90°, and forearm and wrist in a neutral position, and will perform three consecutive tests. The best of these measurements will be recorded in kilograms.

CONTACTS AND LOCATIONS:
Overall Officials: Ümit DÜNDAR, Profesor, Principal Investigator — AFYONKARAHİSAR HEALTH SCİENCES UNİVERSITY
Locations (2):
- Turkey (Türkiye) (2):
  - Afyonkarahisar Health Science University, Afyonkarahisar
  - Afyonkarahisar Health Sciences Unıversity, Afyonkarahisar

REFERENCES:
- [Background] Ashour AA, Yehia RM, ElMeligie MM, Hanafy AF. Effectiveness of high intensity laser therapy on pain, grip strength and median nerve conductivity in pregnant women with carpal tunnel syndrome: A randomized controlled trial. J Hand Ther. 2023 Jul-Sep;36(3):536-545. doi: 10.1016/j.jht.2022.03.005. Epub 2022 Jul 8. PMID 35817691
- [Background] Yigit F, Ordahan B. Effects of high-intensity laser therapy on pain, functional status, hand grip strength, and median nerve cross-sectional area by ultrasonography in patients with carpal tunnel syndrome. Lasers Med Sci. 2023 Oct 31;38(1):248. doi: 10.1007/s10103-023-03913-z. PMID 37906312
- [Background] Ezzati K, Laakso EL, Saberi A, Yousefzadeh Chabok S, Nasiri E, Bakhshayesh Eghbali B. A comparative study of the dose-dependent effects of low level and high intensity photobiomodulation (laser) therapy on pain and electrophysiological parameters in patients with carpal tunnel syndrome. Eur J Phys Rehabil Med. 2020 Dec;56(6):733-740. doi: 10.23736/S1973-9087.19.05835-0. Epub 2019 Nov 18. PMID 31742366
- See also: Effectiveness of high intensity laser therapy on pain, grip strength and median nerve conductivity in pregnant women with carpal tunnel syndrome: A randomized controlled trial — https://pubmed.ncbi.nlm.nih.gov/35817691/
- See also: Effects of high-intensity laser therapy on pain, functional status, hand grip strength, and median nerve cross-sectional area by ultrasonography in patients with carpal tunnel syndrome — https://pubmed.ncbi.nlm.nih.gov/37906312/
- See also: A comparative study of the dose-dependent effects of low level and high intensity photobiomodulation (laser) therapy on pain and electrophysiological parameters in patients with carpal tunnel syndrome — https://pubmed.ncbi.nlm.nih.gov/31742366/